CLINICAL TRIAL: NCT03325751
Title: Non-inferiority Study for Visual Field Mean Defect Estimation Using Sequentially Optimized Reconstruction Strategy (SORS) With an OCTOPUS 900 Perimeter on Healthy and Glaucoma Subjects
Brief Title: Visual Field Defect Estimation Using Sequentially Optimized Reconstruction Strategy on Healthy and Glaucoma Subjects
Status: Completed | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: University of Bern (Other)
Responsible Party: Sponsor
Other Study IDs: 2017-01540
Record Dates: First submitted 2017-10-25; First posted 2017-10-30 (Actual); Last update posted 2020-01-09 (Actual); Status verified 2020-01

CONDITIONS: Glaucoma, Open-Angle
MeSH Terms: conditions — Glaucoma, Open-Angle | interventions — Visual Fields

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy subjects
  Interventions: Diagnostic Test: Visual field testing
- Glaucoma subjects: Patients with primary open-angle-, pseudoexfoliation- or primary angle-closure glaucoma
  Interventions: Diagnostic Test: Visual field testing

INTERVENTIONS:
Diagnostic Test: Visual field testing — Standard Automated Perimetry using a perimeter is one of the most commonly used techniques for measuring perceived visual ability of a subject. For a given eye, it provides quantitative measurements of visual function represented as a 2D spatial visual field map. It is of great clinical importance for diagnosing and monitoring glaucoma and detecting neurological conditions.

SUMMARY:
Perimetry is a well-established method that is used to measure the visual field functions of humans. Commercially available products, such as the OCTOPUS 900 (Haag-Streit AG, Koeniz, Switzerland), are commonly used for assessing the visual field. Such devices are of critical value for patients suffering of glaucoma and neuro-ophthalmic conditions. The operating principle is to sequentially present light stimuli of different intensity at different locations within the visual field in an automatic way. Algorithms that select what locations and intensities to present over time are called strategies. These have the goal to provide both a fast and accurate estimation of the visual field function.

Recently, new strategies were developed that are faster and equally accurate as the strategies used today. The technological advancement of these new methods lies primarily in the ability to estimate location sensitivities without observing them directly but by leveraging previously queried locations. For this the investigators plan to implement the next generation of perimetry strategies into an OCTOPUS 900 and to test it in healthy subjects and glaucoma patients.

ELIGIBILITY:
Inclusion Criteria:

* Cataract yes or no
* Age range 40 - 80 years
* Normal visual field (MD: < +2 dB)
* Refractive error within ±5 dpt. spherical equivalent
* Astigmatism of < -3 dpt.
* Visual acuity of ≥0.3 logMar (decimal ≥0.5)
* Experience in perimetry (history of at least one perimetry examination)
* False positive or negative errors each less than 20% in each examination
* Primary open-angle/ pseudoexfoliation/ primary angle-closure glaucoma
* Early to moderate visual field loss (MD: +2 to +12 dB)
* Written informed consent

Exclusion Criteria:

Exclusion criteria are children (<18 years old), inability to follow the procedure, insufficient knowledge of project language, the history of other ocular diseases than glaucoma or cataract or other conditions that might affect visual field testing (e.g. pituitary lesions, demyelinating diseases).

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy subjects and subjects with Primary open-angle-, pseudoexfoliation- or primary angle-closure glaucoma
Sampling Method: Probability Sample
Enrollment: 103 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-08-02 (Actual); Study Completion 2019-11-01 (Actual)

PRIMARY OUTCOMES:
Non-inferiority estimation quality of mean defect between SORS and dynamic strategy visual field locations | 12 months
  The primary endpoint of this study is the non-inferiority estimation quality of mean defect when using SORS visual field locations as compared to the dynamic strategy visual field locations in healthy subjects and glaucoma patients with early or moderate visual field loss. The non-inferiority margin is defined as a mean defect difference of no more than 0.5 decibel to the dynamic strategy measurement.

CONTACTS AND LOCATIONS:
Overall Officials: René G Höhn, M.D., Principal Investigator — Department of Ophthalmology, Inselspital, University Hospital Bern, University of Bern, Bern, Switzerland
Locations (1):
- Department of Ophthalmology, Inselspital, University Hospital Bern, Bern, Switzerland